CLINICAL TRIAL: NCT01652560
Title: Observational Studies of the Application of Bevacizumab in HER2-negative Breast Cancer Neoadjuvant Chemotherapy
Acronym: BIBC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LiNanlin,Ph.D, Chief Physician,Clinical Professor (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, LiNanlin,Ph.D, Chief Physician,Clinical Professor, The department of Vascular endocrine surgery, Xijing Hospital
Organization: Xijing Hospital (Other)
Other Study IDs: QTDS-01
Record Dates: First submitted 2012-07-21; First posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer; Bevacizumab; Neoadjuvant Chemotherapy; Molecular Targeted Therapy
Keywords: bevacizumab; neoadjuvant chemotherapy; HER2-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- bevacizumab combined neoadjuvant chemotherapy
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: bevacizumab — The patients will be treated with Avastin combined neoadjuvant chemotherapy
  Other Names: Avastin

SUMMARY:
- The purpose of this study is to evaluate the efficacy and safety of the application of bevacizumab combined neoadjuvant chemotherapy in HER2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* HER2-negative breast cancer patients
* Without surgery
* Plans to neoadjuvant chemotherapy

Exclusion Criteria:

* HER2-positive breast cancer patients
* Post-operative patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients of vascular endocrine surgery department in Xijing Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From enrollment to disease progression
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.

SECONDARY OUTCOMES:
overall response | From enrollment to disease progression
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital ， Fourth Military Medical University, Xi'an, Shaanxi, China